CLINICAL TRIAL: NCT04835233
Title: Management of Hypertension in the Early Postpartum Period: Randomized Clinical Trial Comparing Two Antihypertensive Medications
Brief Title: Management of Hypertension in the Early Postpartum: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Rossana Mariana Carvalho de Paiva Marques, MD, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19479
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy-Induced Hypertension in Postpartum; Postpartum Pre-Eclampsia; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Methyldopa

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methyldopa (Experimental): maintaining postpartum the use of methyldopa 250 mg 01 tablet every 8 hours, being able to double the dose depending on pressure levels, up to 15 days postpartum
  Interventions: Drug: Methyldopa 250 MG
- captopril (Active Comparator): postpartum exchange methyldopa for captopril 25 mg 01 tablet every 8 hours, doubling the dose depending on pressure levels, up to 15 days postpartum
  Interventions: Drug: Methyldopa 250 MG

INTERVENTIONS:
Drug: Methyldopa 250 MG — maintaining postpartum the use of methyldopa 250 mg 01 tablet every 8 hours, being able to double the dose depending on pressure levels, up to 15 days postpartum

SUMMARY:
In hypertensive mothers, it is common in clinical practice to substitute methyldopa for another medication, such as captopril, immediately after delivery, which may, as a consequence, cause a rebound effect or an initial lack of blood pressure control until the new medication had a more complete action. Thus, the treatment of hypertension in the puerperium is generally guided by expert opinion and recommendations for guidelines, based on non-robust evidence. OBJECTIVE: To evaluate the control of blood pressure in postpartum women with hypertensive syndromes during pregnancy with the maintenance of the continued use of previously used methyldopa compared to switching from antihypertensive regimen to the use of captopril. METHOD: Randomized, double-blind, drug controlled clinical trial. EXPECTED RESULT: better pressure control with the continued use of methyldopa.

DETAILED DESCRIPTION:
Objective: To evaluate blood pressure control during the immediate postpartum in hypertensive women who had used methyldopa during pregnancy, comparing continuation of that drug with switching it for captopril. Methods: A single-blind, randomized clinical trial involving 180 postpartum women with arterial hypertension who had previously used methyldopa during pregnancy at a minimum dose of 750 mg/day for at least one week prior to delivery. Following delivery, the patients were randomized either to continue with methyldopa (minimum dose 250 mg, three times a day) (methyldopa group, n=90) or to switch to captopril (at an initial dose of 25 mg, three times a day) (captopril group, n=90). Logistic regression will be used to compare the groups regarding the potential to maintain blood pressure below 140/90 mmHg at over 50% of measurements postpartum.

ELIGIBILITY:
Inclusion Criteria:

* puerpera;
* hypertensive;
* use of methyldopa during pregnancy at a minimum dose of 750 mg / day, for at least 07 days before delivery

Exclusion Criteria:

* Use of other antihypertensive medications or illicit drugs that may interfere with maternal hemodynamics, and / or Contraindications to the use of captopril or methyldopa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Values of blood pressure (systolic blood pressure) | every 4 hours immediately after the use of medication until hospital discharge
  systolic blood pressure values in mmHg (millimeters of mercury) after starting postpartum medication
Values of blood pressure (dyastolic blood pressure) | every 24 hours immediately after the use of medication until hospital discharge
  diastolic blood pressure values in mmHg (millimeters of mercury) after starting postpartum medication
Values of blood pressure ( mean arterial pressure) | every 4 hours immediately after the use of medication until hospital discharge
  mean blood pressure values in mmHg (millimeters of mercury) after starting postpartum medication
Values of heart rate | every 4 hours immediately after the use of medication until hospital discharge
  values of heart rate bpm (beat per minute) after starting postpartum medication
Frequency of hypertensive peaks | every 4 hours immediately after the use of medication until hospital discharge
  numbers of hypertensive peaks (Systolic Blood Pressure ≥160 mmHg and / or Diastolic Blood Pressure ≥ 110 mmHg) after starting postpartum medication

SECONDARY OUTCOMES:
Profile of the following laboratory tests ( protein urinary) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the days of puerperium: urinary protein / creatinine (P / C) ratio (measured in mg / dL). Values greater than 300mg/dL of protein in 24h are indicative of pre-eclampsia.
Profile of the following laboratory tests ( urea) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: urea ( blood dosage) measure of value ( mg/dL)
Profile of the following laboratory tests (creatinine) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: creatinine ( blood dosage) measure of value ( mg/dL)
Profile of the following laboratory tests (DHL) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: lactic dehydrogenase -DHL ( blood dosage) measure of value ( UI/L)
Profile of the following laboratory tests (uric acid) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: uric acid (blood dosage) measure of value mg/dL
Profile of the following laboratory tests aspartate transferase (AST)) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: aspartate transferase (blood dosage) measure of value U/L
Profile of the following laboratory tests alanine transferase (ALT) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: alanine transferase (ALT) (blood dosage) measure of value U/L
Profile of the following laboratory tests (total bilirubins, direct and indirect ) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: total bilirubins, direct and indirect (blood dosage)- measure of value U/L
Profile of the following laboratory tests (platelets) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: platelets/ µL (blood dosage)
Profile of the following laboratory tests (glomerular filtration rate) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: calculated by formula Modification of Diet Disease (MDRD) or Chronic Kidney Disease Epidemiology Collaboration ( CKD-EPI), obtained by the site: http://mdrd.com/
Profile of the following laboratory tests (sodium, potassium and chlorine) on admission and their evolution during the puerperium | the first before delivery and the next every 24 hours after delivery until the normalization of the values
  Profile of the following laboratory tests on admission and their evolution during the puerperium: sodium, potassium and chlorine - measure of value (mEq/L)
Days of hospital stay after delivery until blood pressure control | number of days (24 hours) from postpartum hospitalization until normalization of blood pressure
  Days of hospital stay after delivery until blood pressure control (more than 50% of blood pressure measurements less than or equal to 140 x 90 mmHg)
Need for drug use for hypertensive peak ( yes or no) | every 4 hours immediately after the use of medication until hospital discharge
  Clonidine was the drug of choice in the study. The hypertensive peak was considered to be greater than or equal to systolic pressure 160 mmHg and / or diastolic pressure greater than or equal to 110 mmHg.
Need to associate another hypotensive drug to control blood pressure ( yes or no) | immediately after the use of medication until hospital discharge
  Need to associate another hypotensive drug to control blood pressure until blood pressure control (more than 50% of blood pressure measurements less than or equal to 140 x 90 mmHg)
use of analgesic and anti-inflammatory ( yes or no) | number of doses in 24 hours for postpartum analgesia
  need for analgesic and anti-inflammatory use and the amount used (number of doses)
Use of antihypertensive drugs at the time of hospital discharge ( yes or no) | immediately after discharge from the hospital up to 15 days after delivery
  patient was discharged using antihypertensive medication
Frequency of adverse effects most often described with medications ( yes or no) | immediately after the use of medication until hospital discharge
  numbers of adverse effects most often described with medications: drowsiness, headache, dizziness, orthostatic hypotension, nausea, vomiting, diarrhea, dry mouth, dry cough, skin rashes, itching, arthralgia, skin lesions, dysgeusia, angioedema
maternal complicatios ( yes or no) | immediately after the use of medication until hospital discharge
  maternal complications (eclampsia, HELLP syndrome, impending eclampsia, oliguria, puerperal complications and maternal death) and complications related to hypertensive peaks (stroke, acute myocardial infarction and acute lung edema)
satisfactory breastfeeding | immediately after the use of medication until hospital discharge
  satisfactory, unsatisfactory and with difficulty reported by the mother
degree of maternal satisfaction with medication | immediately after the use of medication until hospital discharge
  I hated it, I didn't like it, indifferent, I liked it, I loved it (scale of faces)
Postpartum depression | immediately after the use of medication until return for evaluation of the patient 15 days after delivery
  Edinburgh Postpartum Depression Scale (EPDS)
Neonatal outcomes ( bradycardia) -yes or no | immediately after the use of medication until hospital discharge
  bradycardia( below 100 beats per minute of the newborn)
Neonatal outcomes ( hypoglycemia) -yes or no | immediately after the use of medication until hospital discharge
  blood glucose below < 45 mg/dL
Neonatal outcomes (Hypothermia) -yes or no | immediately after the use of medication until hospital discharge
  Hypothermia below 36,5 degree celsius
Neonatal outcomes (comorbidity) -yes or no | immediately after the use of medication until hospital discharge
  Some unfavorable clinical condition of the newborn (comorbidity)
Neonatal outcomes (hypotension) -yes or no | immediately after the use of medication until hospital discharge
  mean arterial pressure (mmHg) below gestational age (weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Telis Araujo, PhD, Principal Investigator — Federal University of Paraíba; Luiz Aparecido Bortolotto, PhD, Principal Investigator — FMUSP
Locations (1):
- UFPB Paraíba Federal University, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No